CLINICAL TRIAL: NCT07335276
Title: Enhancing Operational Readiness With Digital Self-Managed Cognitive Behavioral Therapy for Insomnia (CBTI): A Pilot Randomized Controlled Trial for Service Members
Brief Title: Enhancing Operational Readiness With Digital Self-Managed Cognitive Behavioral Therapy for Insomnia (CBTI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: TriService Nursing Research Program (Funder) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11207-N25-D03
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Insomnia; Depression - Major Depressive Disorder; PTSD
Keywords: Insomnia; Service Members; Cognitive Behavioral Therapy for Insomnia; Digital Application
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Study design is a prospective, randomized controlled trial with two arms (intervention and wait list control).
Masking Description: All study participants will complete initial study questionnaires and sleep diary data for one week. At one week study participants will be randomized into groups. At this time the study will be unblinded to provide instructions on the intervention and to follow up with participants for questionnaire completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital App CBTI (Experimental): Participants will use a digital app for self-directed CBTI for five weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Waitlist Control (No Intervention): This group will be placed on a waitlist control group until the follow up period is complete.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — This intervention will be delivered via a smart phone app
  Arms: Digital App CBTI

SUMMARY:
The goal of this pilot clinical trial is to evaluate the effectiveness and delivery method of a CBTI self-managed digital mobile application in service members.

The main questions it aims to answer are:

RQ1. Will the delivery of CBTI via a self-managed mobile application over five weeks improve sleep outcomes for service members?

RQ2. Will the delivery of CBTI via a self-managed mobile application over five weeks improve secondary outcomes (sleep-related impairment, depression, PTSD symptoms, and quality of life) for service members?

DETAILED DESCRIPTION:
Participants enrolled in this trial will:

* Week 1: Complete a series of questionnaires (approximately 15 minutes) & complete a daily sleep diary for one week (three minutes each morning).
* Weeks 2-6: Participate in one of two groups that are randomly assigned:
* Group 1: Starts use of the smart phone app with treatment for insomnia for five weeks. Each day during weeks 2-6 you will complete a daily sleep diary on the app and review individual sleep treatment recommendations (total of 5 minutes each morning).

OR

* Group 2: Will wait for five weeks
* End of Week 6: Both Group 1 & Group 2 will complete a series of questionnaires (approximately 15 minutes), & complete a daily sleep diary for one week (three minutes each morning).
* Week 10: Both Group 1 & Group 2 will complete a series of questionnaires (approximately 15 minutes) about insomnia symptoms, any sleep related impaired function, depression symptoms, post-traumatic stress disorder symptoms, and quality of life. Participants randomized to the wait list will be contacted to provide information and support on how to use the smart phone app for treatment with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty, Reservist, Army National Guard
* Ages 18-55 years
* Own a smart phone
* Internet access

Exclusion Criteria:

* Insomnia Severity Score > or equal to 10
* PHQ-8 score <20
* Untreated sleep disorders (sleep apnea, narcolepsy, parasomnias)
* Pregnancy
* Working rotating Shifts
* Caring for a newborn <3 months old
* Currently receiving cognitive behavioral therapy for insomnia
* Received cognitive behavioral therapy for insomnia in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-10-02 (Estimated); Study Completion 2028-10-02 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | Baseline, Six Weeks, Nine Weeks
  Insomnia severity will be measured with the Insomnia Severity Index (ISI). The ISI is a seven-item self-report questionnaire assessing the nature, severity, and impact of insomnia symptoms in the past 2 weeks. Items are rated on scales from 0 - 4 (none-severe). Item ratings are summed to get a total score, with higher scores reflecting greater insomnia severity (0-7 = no clinically significant insomnia, 8-14 = subthreshold insomnia, 15-21 = clinically significant insomnia -moderate, 22-28 = clinically significant insomnia - severe).

SECONDARY OUTCOMES:
Consensus Sleep Diary | Baseline, Six Weeks
  Subjective sleep measures will be captured using the Consensus Sleep Diary (CSD). The CSD is a nine-item tool which provides participant reported daily sleep patterns and sleep outcome measures. The CSD was developed by leading sleep experts in an effort to create a standardized sleep diary for clinicians and researchers. Sleep diaries have been regarded as a gold standard for subjective sleep assessment, and are viewed by sleep experts as a useful methodology for prospective self-monitoring of sleep for individuals with insomnia. Through simple questions delivered via the Insomnia Coach app, participants are asked to report daytime napping, bedtime, time attempted to fall asleep, sleep onset latency (SOL), number of awakenings (NOA), wake after sleep onset (WASO), total sleep time (TST), time of awakening, sleep efficiency (SE), and sleep quality using a 5-point scale from 1-5 (1 = "very poor," 2 = "poor," 3 = "fair," 4 = "good," 5 = "very good").
PROMIS Sleep-Related Impairment 8a | Baseline, Six Weeks, Nine Weeks
  The PROMIS Sleep-Related Impairment 8a (PROMIS-SRI 8a) is an 8-item self-report measure assesses daytime sleep-related impairment (SRI) over the past seven days. The PROMIS Sleep-Related Impairment 8a is the short form of the PROMIS-SRI 16. Each item has five response options ranging from 1- 5 (1 = "not at all," 2 = "a little bit," 3 = "somewhat," 4 = "quite a bit," 5 = "very much"). Higher scores indicating greater daytime function disturbances (range 0-40). Item ratings are summed to compute a raw score, which is converted to a standardized T score using conversion tables published on the Patient-Reported Outcomes Measurement Information System (PROMIS) website (nihpromis.org).
The Post Traumatic Stress Disorder Checklist-Military Version (PCL-M) | Baseline, Six Weeks, Ten Weeks
  The Post Traumatic Stress Disorder Checklist-Military Version (PCL-M) is a self-report questionnaire designed to assess the symptoms of PTSD in which 17 items correspond to the Diagnostic and Statistical Manual of Mental Disorders PTSD criteria. Items one through five correspond to re-experiencing symptoms, items five and six correspond to avoidance symptoms, items eight through twelve correspond to numbing symptoms, and items thirteen through seventeen correspond to hyperarousal symptoms. Individuals are asked to endorse the level of distress with each symptom over the last 30 days. Items are scored on a five-point Likert scale with 1 = "not at all" to 5 = "extremely." A total symptom severity score is obtained (range 17-85), with higher scores indicating higher PTSD symptoms and scores greater than 50 indicating a high likelihood of PTSD diagnosis.
The Patient Health Questionnaire-8 (PHQ-8) | Baseline, Six Weeks, Nine Weeks
  The Patient Health Questionnaire-8 (PHQ-8) is an eight item self-report questionnaire used to examine depression severity with similar psychometric properties of the PHQ-9. The PHQ-8 omits the final question of the PHQ-9 regarding suicide as the electronic delivery of the instruments may not provide timely clinical response to a positive endorsement of this question. Individuals are asked to endorse the level of distress with each symptom on the PHQ-9 in the last two weeks. A four-point Likert scale with 0 = "not at all," 1 = "several days," 2 = "more than half the days," and 3 = "nearly every day" is used. A total symptom severity score is obtained (range 0-24). Severity of depression is scored as follows: 0-4 no significant depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-24 severe depression. Scores greater than ten indicate a high likelihood of depression.
RAND-36 Item Short Form Survey | Baseline, Six Weeks, Ten Weeks
  The RAND-36 Item Short Form Survey (RAND-36) is a health-related quality of life questionnaire that assesses how health impacts on an individual's ability to function & their perceived well-being in physical, mental and social domains of life. The RAND-36 includes a total of 36 items which includes eight domains representing aspects of health and quality of life: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Each domain includes either Likert type questions (with either 1-5 or 1-3 scales) and binary yes/no questions. The 36 items are grouped by the eight domains and each domain has a profile score (range 0-100). Higher scores within each domain indicate better health, higher quality of life, and less functional limitation.

IPD SHARING:
Plan to Share IPD: Undecided
Participant de-identified data sharing has not been determined at this point in time. Considerations include this data is DoD data and since the study has not started, it is unknown how much data or the quality of the data that will be obtained.